CLINICAL TRIAL: NCT03063333
Title: Long-term Effect of Hypnosis in Spinal Cord Injury Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Head of project stopped
Sponsor: Lone Knudsen, MSc Psych, PhD (Other)
Responsible Party: Sponsor-Investigator, Lone Knudsen, MSc Psych, PhD, Psychologist, Central Jutland Regional Hospital
Organization: Central Jutland Regional Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 240929
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; hypnosis; pain; pain catastrophizing; coping
MeSH Terms: conditions — Spinal Cord Injuries; Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with three arms: coping-oriented hypnosis, neutral hypnosis, no hypnosis
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coping-oriented hypnosis (Experimental)
  Interventions: Other: Coping-oriented hypnosis
- Neutral hypnosis (Placebo Comparator)
  Interventions: Other: Neutral hypnosis
- current treatment only (No Intervention)

INTERVENTIONS:
Other: Coping-oriented hypnosis — Hypnosis using coping-oriented suggestions based on reversal of statements from the pain catastrophizing scale plus current treatment.
  Arms: Coping-oriented hypnosis
Other: Neutral hypnosis — Hypnosis using neutral suggestions plus current treatment
  Arms: Neutral hypnosis

SUMMARY:
Coping-oriented hypnotic suggestions aimed at reducing pain catastrophizing was shown to reduce pain in people with chronic tension-type headache and experimental pain in healthy volunteers during hypnosis (Kjøgx et al., 2016). However, the duration of the effect on pain post-hypnosis is unknown.

The aim is to investigate the durational effect of a single session of coping-oriented hypnotic suggestions on chronic pain in patients with spinal cord injury. If effective for a longer period post-hypnosis, this form of hypnosis may provide an alternative to medicine or may be used in conjunction with lower medicine dosages.

Methods: 75 patients with spinal cord injury and pain is randomized into one of three conditions; coping-oriented hypnosis plus current treatment, neutral hypnosis plus current treatment or current treatment only. Pain intensity, coping strategies, pain catastrophizing, anxiety and depression is assessed before intervention and over a period of 14 days post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (tetraplegia or paraplegia) with some preservation of hand functioning
* Baseline pain level of ≥ 3 on a Numeric Rating Scale (NRS; 0-10 where 10 is extremely severe pain)
* Pain duration of at least 8 weeks.

Exclusion Criteria:

* Severe mental or psychiatric illness
* Substance abuse (drugs, alcohol or medicine)
* Lack of ability to cooperate during the experiment
* Severe high cervical lesions
* Severe autonomic dysautonomia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | For 14 days post-intervention
  NRS (0-10)
Coping | For 14 days post-intervention
  Coping strategies questionnaire

SECONDARY OUTCOMES:
Pain catastrophizing | For 14 days post-intervention
  Pain catastrophizing scale
Pain impact on mood, sleep and daily activities | For 14 days post-intervention
  NRS (0-10)
Anxiety | For 14 days post-intervention
  Hospital Anxiety and Depression Scale
Depression | For 14 days post-intervention
  Hospital Anxiety and Depression Scale
Global impression of change | For 14 days post-intervention
  Global impression of change scale

OTHER OUTCOMES:
Side effects | For 14 days post-intervention
  patient report

CONTACTS AND LOCATIONS:
Overall Officials: Helge Kasch, MD, PhD, Study Chair — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Spinal Cord Injury Centre of Western Denmark, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kjogx H, Kasch H, Zachariae R, Svensson P, Jensen TS, Vase L. Experimental manipulations of pain catastrophizing influence pain levels in patients with chronic pain and healthy volunteers. Pain. 2016 Jun;157(6):1287-1296. doi: 10.1097/j.pain.0000000000000519. PMID 26871534